CLINICAL TRIAL: NCT02901210
Title: A Modified Technique to Facilitate Pealing of the Rectal Mucosa in Delorme Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasser Mohamed Abdel-samii (Other)
Responsible Party: Sponsor-Investigator, Yasser Mohamed Abdel-samii, Lecturer of general surgery., Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006379
Record Dates: First submitted 2016-07-14; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Rectal Prolapse
Keywords: Recta prolapse; Intraoperative bleeding; mucosal cauterization
MeSH Terms: conditions — Rectal Prolapse; Blood Loss, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Modified Delorme (Experimental): Modified technique for delorme procedure done in mild to moderate rectal prolapse as the investigator destroy use the electrocautery to peal the mucosa with less intraoperative bleeding ,avoiding stripping of the mucosa done in classic delorme that induce major bleeding intraoperative .
  Interventions: Procedure: Modified delorme procedure

INTERVENTIONS:
Procedure: Modified delorme procedure

SUMMARY:
The aim of this study is to evaluate the investigator new modification for delorme procedure in patients with rectal prolapse , assessing intra-operative morbidity and recurrence rate .

DETAILED DESCRIPTION:
In classic delorme operation stripping of the mucosa done and this is associated with extensive bleeding in addition to the time consumed in this step.the new modification done by the investigator replace this step with another associated with less intraoperative bleeding and not time consuming.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate rectal prolapse
* Singed informed consent.

Exclusion Criteria:

* Huge rectal prolapse .
* Recurrent rectal prolapse

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Recurrence rate assessed in this modified technique | One year follow up post operative
intraoperative bleeding measured in this modified technique | one year follow up post operative.

IPD SHARING:
Plan to Share IPD: Undecided